CLINICAL TRIAL: NCT01650792
Title: CHADSS: Chagas Disease Scan Study
Brief Title: Clinical Assessment, Neuroimaging and Immunomarkers in Chagas Disease Study (CLINICS)
Acronym: CLINICS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Bahia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jamary Oliveira-Filho, Associate Professor, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS064905 (NIH); R01NS064905 (NIH)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chagas Disease With Heart Failure
Keywords: Chagas disease; Heart failure; Stroke; Dementia
MeSH Terms: conditions — Chagas Disease; Heart Failure; Stroke; Dementia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin 300mg per day for 7 days in patients with HITS on transcranial Doppler monitorization
  Interventions: Drug: Aspirin
- Best medical treatment (No Intervention): Best medical treatment including drugs for heart failure and hypertension will be given to both groups.

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin

SUMMARY:
The main purpose of the study is to determine noninvasive markers of brain involvement in Chagas disease. In a subgroup of patients with high intensity transient signals (HITS) on transcranial Doppler monitorization, the investigators aim to determine the efficacy and safety of aspirin in preventing microembolization in patients with no previous history of stroke. Specific aims are listed bellow:

(1) to establish brain magnetic resonance imaging markers of stroke risk in patients with Chagasic heart failure (HF); (2) to determine whether biomarkers can predict stroke risk in patients with Chagasic HF; and (3) to evaluate the efficacy of antiplatelet treatment in decreasing microembolization rate in patients with Chagasic HF.

DETAILED DESCRIPTION:
Stroke is an enormous international public health concern, particularly in the developing world where there are limited resources available to provide for an aging population. One of the main contributors to stroke incidence is the highly prevalent Chagas disease, a parasitic infection affecting an estimated 18 million individuals and a major cause of heart failure in Latin America. Chagas disease conveys stroke risk through two established mechanisms: structural cardiac disease and chronic inflammation. Although inflammation is associated with an increased risk of ischemic stroke and poorer outcome, its role has been largely linked to atherogenesis. Chronic inflammation can result in endothelial dysfunction and stimulate the hemostatic system, increasing systemic fibrin production and platelet activation. Brain atrophy has also been associated with chronic inflammation. Adults, young and old, who develop a secondary cardiomyopathy from Chagas are therefore at higher risk of cardioembolism and neurodegeneration. Stroke patients usually survive, but can be left with significant disability affecting their health status, productivity, and quality of life. These factors impact caregivers as well. Thus, the social and economic consequences of stroke are vast. During our R21 planning grant period, we were able to establish a collaborative infrastructure between the research groups in Brazil and the United States and collect preliminary data. We found an association between Chagas disease and stroke that was independent of cardiomyopathy. Cognitive impairment and brain atrophy were also associated with Chagas disease independently of cardiomyopathy. Biomarkers orosomucoid, neprilysin, interleukin-6 (IL-6) and matrix metalloproteinase-9 (MMP-9) were identified as diagnostic and therapeutic targets in Chagas disease. As part of this phase, we will address three specific aims: (1) to establish brain magnetic resonance imaging markers of stroke risk in patients with Chagasic congestive heart failure (CM); (2) to determine whether biomarkers can predict stroke risk in patients with Chagasic CM; and (3) to evaluate the efficacy of antiplatelet treatment in decreasing microembolization rate in patients with Chagasic CM. The long-term goal of this project is to establish non-invasive methods of stroke risk stratification and prediction of stroke outcome in patients with Chagas disease. This work will also facilitate the development of novel anti-trypanosomal, anti-inflammatory, and antithrombotic strategies for stroke prevention and management in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure according to Framingham criteria
* Informed consent
* Age 18 years or above

Exclusion Criteria:

* Patients with a history of an untreated malignancy (except local skin cancers)
* Ischemic stroke (determined using the Questionnaire for Verifying Stroke-Free Status (QVSFS)
* Patients on renal dialysis or with end-stage hepatic dysfunction
* Acute infection/inflammation (Temperature > 101.5 F, and/or WBC> 15, 000)
* Inability to obtain informed consent from patient or next of kin
* Anticoagulant use (warfarin or heparin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Brain magnetic resonance imaging lesions | Baseline cross-sectional data
  Primary hypothesis is that silent brain infarcts, brain atrophy and white matter disease will be more common in patients with Chagas disease heart failure when compared to other etiologies of heart failure.
Biomarkers | Baseline cross-sectional data
  Primary hypothesis is that serum biomarkers orosomucoid, neprilysin, interleukin-6 and matrix metalloproteinase-9 will be increased in Chagas disease heart failure when compared to other etiologies of heart failure
Proportion of high intensity transient signals on transcranial Doppler monitorization | One week
  Primary hypothesis is that the proportion of patients with high intensity transient signals (HITS) on one-hour transcranial Doppler monitorization after one-week treatment with 300mg aspirin and best medical treatment will be less when compared with best medical treatment without aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Jamary Oliveira-Filho, MD, PhD, Principal Investigator — Associate Professor, Federal University of Bahia
Locations (1):
- Hospital Universitario Professor Edgard Santos, Salvador, Estado de Bahia, Brazil